# Graphic Messages to Prevent E-Cigarette Use Among Latino and African American Adolescents: A Randomized Controlled Trial

# **Informed Consent Form**

NCT04899999

Date: 6/18/2021

Date: 6/18/2021



Date: XX/XX/XXXX

## Information Sheet

## Dear Parent(s)/Caregiver(s),

This information sheet explains why we are doing this research, and what it will involve. Please take time to read this information carefully together with your adolescent. Please contact the research team (contact below) if there is anything that is not clear or if you would like more information. Thank you for reading this document.

**Project title:** Graphic messages to prevent e-cigarette use among Latino and African American adolescents: A randomized controlled trial

Principal Investigator: Dr. Francisco Cartujano

#### What is this study about?

Vaping products have completely transformed the landscape of nicotine use in adolescents and is now two to three times more common among adolescents than adults. Although initially marketed as an effective mean for smoking cessation, recent research shows that exposure to nicotine during adolescence and young adulthood is not only associated with increased rates of use of other substances, but also has long-term effects on the developing brain. Therefore, there is an urgent need to prevent vaping among adolescents. However, one of the limitations of the existing research on adolescents and vaping-use is the lack of representation of Latino and African Americans. This leaves a substantial gap in communication research for vaping prevention among racial and ethnic groups. As the adolescent vaping epidemic continues to grow, there is an urgent need to develop, test, and implement messages and communication channels for vaping prevention. This study aims to determine if graphic messages prevent future vaping use among African American and Latino adolescents.

### How will my adolescent be involved?

If your adolescent decides to take part in this study, your adolescent will be asked to complete an online survey via REDCap, a secure web-based system. The online survey will collect sociodemographic characteristics and susceptibility to future vaping use. While completing the survey, your adolescent will be randomized to one of four groups: 1) Financial reward graphic message, 2) Health reward graphic message, 3) Self-efficacy graphic message, or 4) Social norms graphic message. In each of these groups, your adolescent will receive one image via REDCap that targets vaping use. Your adolescent will be instructed to look at this image and caption for as long as they wish and will be given a brief survey to complete afterwards that will

RSRB Approval Date: 6/18/2021

assess for likelihood of future vaping use. Participating in this study will take approximately 45 minutes. As a compensation of the time and effort, your adolescent will receive \$25 gift card at the end of the assessment. We estimate that approximately 360 adolescents will take part in this research study.

#### How will your privacy be protected?

In order to collect study information, we have to get your permission and your adolescent's assent to participate in the study. We will use 1) a baseline assessment on sociodemographic characteristics (age, gender, race, ethnicity, etc.) and susceptibility to future vaping, and 2) their post-exposure (to the graphic messages) reactions on likelihood of future vaping. Each subject whose data is collected will be assigned a unique study number. Only the study number will be included in the data collection tool, data analysis tools, and potential publications. Any sensitive data will not be collected.

#### Use of text messaging communication for research

Text messages by mobile/cell phones are a common form of communication. This research study involves sending your adolescent one text message only with the link to complete the online survey and a unique username and password to access the survey.

#### Who do I speak to if I have questions about this research?

If you would like more information regarding the research, please contact Dr. Francisco Cartujano by email at <a href="mailto:Francisco\_Cartujano@URMC.Rochester.Edu">Francisco\_Cartujano@URMC.Rochester.Edu</a> or telephone at 585-287-4539.

Please contact the University of Rochester Research Subjects Review Board at 265 Crittenden Blvd., CU 420628, Rochester, NY 14642, telephone 585-276-0005 or 877-449-4441 for the following reasons:

- You wish to talk to someone other than the research staff about your rights as a research subject;
- To voice concerns about the research;
- To provide input concerning the research process;
  In the event the study staff could not be reached.

#### Can you change your mind?

You and/or your adolescent have the right to withdraw from the research at any time by contacting the research team.

Thank you very much for your time.

Regards,

#### Francisco Cartujano, MD

Research Assistant Professor Department of Public Health Sciences University of Rochester Medical Center

# Chiamaka Azogini, MS4

Student Research Fellow M.D. Candidate | Class of 2022 University of Rochester School of Medicine and Dentistry

RSRB Approval Date: 6/18/2021